CLINICAL TRIAL: NCT04600609
Title: Examining the Experiences of Children With Blood Disorders
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ayesha Zia, Associate Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0772
Record Dates: First submitted 2020-09-22; First posted 2020-10-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Blood Disease; Thrombotic Disorder; Venous Thromboembolism; Hemostatic Disorder; Bleeding Disorder
MeSH Terms: conditions — Hematologic Diseases; Thrombosis; Venous Thromboembolism; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 3-phase mixed methods study design. A literature review (Phase 1) has been completed to determine the areas of exploration and to identify challenges faced and the impact of the blood disorder on pediatric patients. Based on Phase 1, Phases 2 and 3, as proposed in this study, will be completed and will include interviews of patients diagnosed with bleeding and thrombotic disorders (phase 2). The interviews will be individual, semi-structured, and consist of open-ended questions to elicit unbiased and in-depth responses to gain an understanding of participant's perspectives on themes predetermined in the study design phase.

DETAILED DESCRIPTION:
The purpose of this study is to explore the experiences of pediatric patients with blood disorders, specifically thrombotic, including venous thromboembolism (VTE), and hemostatic or bleeding disorders. The information gleaned from this study will help identify specific challenges faced by patients with hemostatic and thrombotic disorders - information that is necessary to develop impactful, evidence-based solutions to support patients with hemostatic and thrombotic disorders cope with the physical, emotional, and psychological impact of blood disorders. Participants with blood disorders in this study will participate in open-ended, semi-structured interviews with a study investigator focusing on the psychosocial experiences of patients with diagnosis and treatment of their underlying disorder and the understanding of their diagnosis. Female participants additionally will be asked questions about the unique effects of heavy menstrual bleeding, either from their underlying blood disorder or secondary to anticoagulation, on similar aspects of the impact of having a blood disorder. Validated questionnaires will be completed to obtain concurrent quantitative data. The interviews will be recorded and transcribed. Participation is complete after the interview has finished; participants will continue to receive standard of care treatment during and beyond the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they are between the ages of 12 and 21 years of age, English speaking and have a formal diagnosis of a hemostatic or thrombotic disorder. For thrombotic disorder patients, an additional eligibility criterion will be to include participants within 1 year of diagnosis.

Exclusion Criteria:

* Patients will be excluded if they do not have access to the technology needed to participate in a virtual interview visit (by telephone).

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will include children (defined as persons who have not attained the legal age for consent to treatments or procedures involved in the research, under the applicable law of the jurisdiction in which the research will be conducted), patients (defined as individuals in a clinical setting with whom there is a treatment relationship), and non-English speakers.
  Patients must meet the eligibility criteria in order to participate in this trial.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Effect of blood disorder diagnosis on quality of life will be measured using Pediatric Quality of Life Questionnaire, Menorrhagia Impact Questionnaire, and Godin Physical Activity Questionnaire
Patient confidence assessment | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Patient confidence in managing blood disorder and recognizing emergencies will be assessed using a semi-structured interview with the patient
Quality of care assessment | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Impressions of quality of care received in a specialized bleeding disorders and thrombosis clinic will be assessed using a semi-structured interview with the patient
Implications on the future for the patient with the bleeding disorder | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Patient's reaction to the diagnosis and its impact on their future will be assessed using a semi-structured interview with the patient

SECONDARY OUTCOMES:
Depression screening | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Screening completed using PHQ-9 questionnaire
Quality of life screening | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Screening completed using Peds QOL questionnaire
Menorrhagia screening for participants with bleeding disorders | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Screening completed using Menorrhagia impact questionnaire
Dalhousie Dypsnea screening for participants with clots | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Screening completed using Dalhousie Dypsnea questionnaire
Physical activity screening | Within 1 year of diagnosis for clot patients; after formal diagnosis for bleeding disorder patients
  Screening completed using Godin Physical Activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Zia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Parker M, Hannah M, Zia A. "If I wasn't a girl": Experiences of adolescent girls with heavy menstrual bleeding and inherited bleeding disorders. Res Pract Thromb Haemost. 2022 May 30;6(4):e12727. doi: 10.1002/rth2.12727. eCollection 2022 May. PMID 35664533